CLINICAL TRIAL: NCT02939027
Title: Study of Electronic Brachytherapy for Cutaneous Basal Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCCBrachy
Record Dates: First submitted 2016-10-13; First posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Carcinoma, Basal Cell
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): For the first 20 patients, a total dose of 36.6 Gy is planned over 6 fractions of 6.1 Gy, given 2 days week, 3 weeks or lees at least 2 days apart each fraction.
  Interventions: Device: Electronic Brachytherapy (6,1 Gy)
- Group 2 (Experimental): For the next 20 patients a total dose of 42 Gy is planned over 6 fractions of 7 Gy, given 2 days week 3 weeks or lees at least 2 days apart each fraction.
  Interventions: Device: Electronic Brachytherapy (7 Gy)

INTERVENTIONS:
Device: Electronic Brachytherapy (6,1 Gy) — A total dose of 36.6 Gy is planned over 6 fractions of 6.1 Gy, given 2 days/week, during 3 weeks or lees, at least 2 days apart each fraction.
  Arms: Group 1
Device: Electronic Brachytherapy (7 Gy) — A total a dose of 42 Gy is planned over 6 fractions of 7 Gy, given 2 days/week during 3 weeks or lees, at least 2 days apart each fraction.
  Arms: Group 2

SUMMARY:
Electronic brachytherapy (EBT) offers an isotope-free radiation therapy modality for the treatment of specific skin lesions, especially non-melanoma skin cancers (NMSC). Within the treatment of NMSC, surgical removal of the lesion is currently the treatment of choice for the majority of cases. However in an estimated 10-15% of NMSC patients, surgery might not be the best treatment option. Location of the tumour in cosmetically sensitive areas, patient comorbidities, old age, use of anti-coagulation etc. might all be reasons to select radiotherapy as first choice of treatment. The objective of ths study will be to determine histologically confirmed clinical efficacy, safety, and usability of Electronic Brachytherapy, an innovative treatment for Basal Cell Carcinoma (BCC).

DETAILED DESCRIPTION:
* Rationale: Electronic brachytherapy (EBT) offers an isotope-free radiation therapy modality for the treatment of specific skin lesions, especially non-melanoma skin cancers (NMSC). Within the treatment of NMSC, surgical removal of the lesion is currently the treatment of choice for the majority of cases. However in an estimated 10-15% of NMSC patients, surgery might not be the best treatment option. Location of the tumour in cosmetically sensitive areas, patient comorbidities, old age, use of anti-coagulation etc. might all be reasons to select radiotherapy as first choice of treatment.
* Objective: To determine histologically confirmed clinical efficacy, safety, and usability of Electronic Brachytherapy, an innovative treatment for Basal Cell Carcinoma (BCC).
* Study design: Prospective, out-patient based, single centre, single treatment modality
* Study population: 40 patients, >18 years old, having at least 1 BCC. Intervention: BCC will be treated with EBT, using low-energy X-rays. Area of the lesion will be evaluated for tumour presence and size before, during and at 2 weeks, 6 weeks and 3 months after treatment. If the patient has more than one BCC, all of them will be treated with Electronic Brachytherapy but only the largest one will be analysed in the study.
* Main study parameters/endpoints: Local control of BCC.
* Secondary parameters: Acute skin toxicity, skin cosmesis, and care giver satisfaction, and patient satisfaction.
* Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients will be exposed to low-energy X-rays. Required site-visits are: 1 pretreatment visits (intake/informed consent and biopsy), 6 treatment visits over the course of 2-3 weeks, 6 control-visits 2 weeks, 6 weeks, 3 months, 6 months, 12 months and 24 months after treatment.
* Patients will also be asked to complete a short questionnaire to evaluate their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥18 years old.
* Estimated life expectancy of ≥5 years
* Histopathologic diagnosis of early and primary Basal Cell Carcinoma (BCC)
* Clinical stage of BCC: T1 or T2 (by AJCC 2010 criteria, see Table 1)
* Histological subtypes: Superficial BCC or nodular BCC
* Maximum diameter of lesion: 20 mm
* Maximum depth of invasion: 4 mm.
* Ability to provide informed consent
* Punch biopsy of primary tumor to depth of reticular dermis

Exclusion Criteria:

* Men or women <18 years old.
* Estimated life expectancy <5 years.
* BCC that was previously treated (ie, recurrent BCC)
* BCC in region adjacent to or overlapping with region of prior radiotherapy
* BCC on irregular surface (ie, target area not flat)
* BCC adjacent to or overlapping with burn or scar
* BCC in area prone to trauma
* BCC in area with compromised lymphatic drainage or vascular supply
* Inflammatory process in target area
* Pregnancy or lactation
* Collagen vascular disease (lupus, scleroderma, rheumatoid arthritis)
* Diabetes that is poorly controlled (Hg A1c >7%)
* Genetic disorder predisposing patient to skin cancers or radiation sensitivity (basal cell nevus syndrome, xeroderma pigmentosum, ataxia telangiectasia mutans)
* Receipt of treatment with another investigational device or drug
* Receipt of drug that will affect biologic response to radiation (radiosensitizer or radioprotector)
* Receipt or plan to receive chemotherapy within 6 weeks of radiation therapy
* High likelihood of protocol non-compliance (in opinion of investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Clinical Response of Electronic Brachytherapy | 2 weeks after treatment
  Response criteria: Complete response (disappearance of tumor), partial response persistence with tumor size reduction), no response (no change in tumor size), tumor progression (increase in tumor size).
Clinical Response of Electronic Brachytherapy | 6 weeks after treatment
  Response criteria: Complete response (disappearance of tumor), partial response persistence with tumor size reduction), no response (no change in tumor size), tumor progression (increase in tumor size).
Clinical Response of Electronic Brachytherapy | 3 months after treatment
  Response criteria: Complete response (disappearance of tumor), partial response persistence with tumor size reduction), no response (no change in tumor size), tumor progression (increase in tumor size).
Clinical Response of Electronic Brachytherapy | 6 months after treatment
  Response criteria: Complete response (disappearance of tumor), partial response persistence with tumor size reduction), no response (no change in tumor size), tumor progression (increase in tumor size).
Clinical Response of Electronic Brachytherapy | 12 months after treatment
  Response criteria: Complete response (disappearance of tumor), partial response persistence with tumor size reduction), no response (no change in tumor size), tumor progression (increase in tumor size).
Clinical Response of Electronic Brachytherapy | 24 months after treatment
  Response criteria: Complete response (disappearance of tumor), partial response persistence with tumor size reduction), no response (no change in tumor size), tumor progression (increase in tumor size).

SECONDARY OUTCOMES:
Patient quality of life | Before treatment and at 3 months post treatment.
  Patient quality of life before and after treatment with Esteya Electronic brachytherapy will be measured using the validated Skindex 16 questionnaire. Patient quality of life will be measured before treatment and at 3 months post treatment.
Rate of grade ≥3-4 adverse events | 2 weeks, 6 weeks, 3 months, 6 months, 12 months and 24 months after treatment.
  The study will use the EORTC-RTOG and Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 for assessing toxicity related to brachytherapy. Grade 4 or higher adverse events will be reported, with the exception of grade 4 radiation dermatitis. Grade 5 radiation dermatitis will be reported.
Caregiver experience (questionnaire) | 3 weeks
  User experience with the Esteya electronic brachytherapy device will be measured using the USE Questionnaire (http://hcibib.org/perlman/question.cgi?form=USE). All users of the device will be asked to fill in one questionnaire after their last use of the treatment device. Only one questionnaire will be filled in per user.

IPD SHARING:
Plan to Share IPD: Undecided